CLINICAL TRIAL: NCT01802749
Title: Multicenter Phase III Randomized Study With Second Line Chemotherapy Plus or Minus Bevacizumab in Patients With Platinum Sensitive Epithelial Ovarian Cancer Recurrence After a Bevacizumab/Chemotherapy First Line
Brief Title: Bevacizumab Beyond Progression in Platinum Sensitive Ovarian Cancer
Acronym: MITO16MANGO2b
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Collaborators: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MITO-16 -MANGO-OV2b; 2012-004362-17 (EudraCT Number); ENGOT-ov 17 (Other: ENGOT)
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Recurrent Ovarian Cancer
Keywords: second line; platinum sensitive; first line bevacizumab; biologic factors; clinical factors
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; Paclitaxel; Carboplatin; liposomal doxorubicin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chemotherapy (Active Comparator): Combination chemotherapy with ONE of the following regimens:
  * PLD-C: Pegylated liposomal doxorubicin 30 mg/m2 + Carboplatin AUC (area under curve) 5 on day 1 every 4 weeks;
  * GEM-C: Gemcitabine 1000 mg/m2 on day 1, 8 every 21 + Carboplatin AUC of 4 on day 1 every 21 days;
  * PAC-C: Paclitaxel 175 mg/m2 on day 1, every 21 + Carboplatin AUC of 5 on day 1 every 21 days.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: pegylated liposomal doxorubicin; Drug: Gemcitabine
- Chemotherapy and bevacizumab (Experimental): Combination chemotherapy AND bevacizumab with ONE of the following regimens:
  * PLD-C: Pegylated liposomal doxorubicin 30 mg/m2 + Carboplatin AUC 5 on day 1 every 4 weeks and Bevacizumab 10 mg/kg i.v. on Day 1 every 2 weeks;
  * GEM-C: Gemcitabine 1000 mg/m2 on day 1, 8 every 21 + Carboplatin AUC of 4 on day 1 every 21 days AND Bevacizumab 15 mg/kg i.v. on Day 1 every 3 weeks;L
  * PAC-C: Paclitaxel 175 mg/m2 on day 1, every 21 + Carboplatin AUC of 5 on day 1 every 21 days AND Bevacizumab 15 mg/kg i.v. on Day 1 every 3 weeks.
  Patients whose disease has not progressed after the initial six cycles of combination treatment will continue bevacizumab, at 15 mg/kg every 3 weeks until disease progression,unacceptable toxicity or patient withdrawn.
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin; Drug: pegylated liposomal doxorubicin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Bevacizumab
  Other Names: Avastin
  Arms: Chemotherapy and bevacizumab
Drug: Paclitaxel
Drug: Carboplatin
Drug: pegylated liposomal doxorubicin
  Other Names: Caelyx
Drug: Gemcitabine

SUMMARY:
Bevacizumab has been found to prolong progression free survival in first line, and more recently, in second line treatment for platinum sensitive ovarian cancer patients who had not received prior treatment with bevacizumab.

Recently reported data suggest that patients with colon cancer who receive bevacizumab in more than one line of therapy (beyond progression) have better results. In ovarian cancer, the role of bevacizumab administered in both first and second-line therapies needs to be defined.

This study aims to evaluate whether administering bevacizumab in combination with chemotherapy in second-line therapy to patients with recurrent ovarian cancer who have received first-line bevacizumab will be more effective than chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥18 years of age.
* Patients with histologically confirmed epithelial ovarian or fallopian tube carcinoma or primary peritoneal carcinoma, including mixed Mullerian Tumours
* Recurrence or progression at least 6 months after the last chemotherapy cycle of a first line carboplatin + paclitaxel chemotherapy including bevacizumab (recurrence or progression might occur either during or after bevacizumab as maintenance)
* Patients can be included if they have a RECIST progression, with either measurable or non-measurable disease
* ECOG (Eastern Cooperative Oncology Group Performance) Status of 0-2.
* Life expectancy of at least 12 weeks.
* Signed informed consent obtained prior to initiation of any study-specific procedures and treatment as confirmation of the patient's awareness and willingness to comply with the study requirements including blood samples for molecular analyses.
* Availability of tumour samples for molecular analyses from primary surgery (mandatory) and secondary surgery (when available)

Exclusion Criteria:

Cancer related

* Ovarian tumours with low malignant potential (i.e. borderline tumours)
* History or evidence of synchronous primary endometrial carcinoma, unless all of the following criteria related to the endometrial carcinoma are met:

  * stage ≤Ia
  * no more than superficial myometrial invasion
  * no lymphovascular invasion
  * not poorly differentiated (grade 3 or papillary serous or clear cell carcinoma).
* Other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix or squamous carcinoma of the skin, or adequately controlled limited basal cell skin cancer.

Prior current or planned treatment:

* More than one previous chemotherapy line
* Previous therapy with other anti-angiogenetic agents different from bevacizumab.
* Any prior radiotherapy to the pelvis or abdomen.
* Surgery (including open biopsy) within 4 weeks prior to the first bevacizumab dose.Current or recent (within 10 days prior to the first study drug dose) use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes (except for line patency, in which case international normalized ratio [INR] must be maintained below 1.5). Post operative prophylaxis with low molecular weight heparin sc is allowed.
* Current or recent (within 30 days of first study dosing) treatment with any other investigational drug.

Laboratory:

* Inadequate bone marrow function: ANC (absolute neutrophil count): <1500/mm3, or platelet count <100,000/mm3 or Haemoglobin <9 g/dl. Patients may be transfused to maintain haemoglobin values ≥9 g/dl.
* Inadequate coagulation parameters:

  * activated partial thromboplastin time (APTT) >1.5 x upper limit of normal (ULN) or
  * INR (international normalized ratio) >1.5
* Inadequate liver function, defined as:

  * serum (total) bilirubin >1.5 x ULN for the institution
  * AST/SGOT or ALT/SGPT > 2.5 x ULN.
* Inadequate renal function, defined as:

  * serum creatinine >2.0 mg/dl or >177 micromol/l
  * urine dipstick for proteinuria >2+. Patients with ≥ 1+ proteinuria at baseline dipstick analysis should undergo a 24-hour urine collection and must demonstrate ≤1g of protein in their 24-hour urine collection.

Prior or concomitant conditions or procedures:

* History or evidence of brain metastases or spinal cord compression.
* Pregnant or lactating females.
* History or evidence of thrombotic or haemorrhagic disorders; including cerebrovascular accident (CVA) / stroke or transient ischemic attack (TIA) or sub-arachnoid haemorrhage within ≤6 months prior to the first study treatment).
* Uncontrolled hypertension (sustained systolic >150 mm Hg and/or diastolic >100 mm Hg despite antihypertensive therapy) or clinically significant (i.e. active) cardiovascular disease, including:
* myocardial infarction or unstable angina within ≤6 months prior to the first study treatment
* New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF)
* serious cardiac arrhythmia requiring medication (with the exception of atrial fibrillation or paroxysmal supraventricular tachycardia)
* peripheral vascular disease ≥grade 3 (i.e. symptomatic and interfering with activities of daily living requiring repair or revision).
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess, or with signs of impending bowel obstruction within 6 months prior to the first study treatment.
* Non-healing wound, ulcer or bone fracture. Patients with granulating incisions healing by secondary intention with no evidence of facial dehiscence or infection are eligible but require three weekly wound examinations.
* Evidence of any other medical conditions (such as psychiatric illness, peptic ulcer, etc.), physical examination or laboratory findings that may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2013-11; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 12 months
  assessed by local Investigator

SECONDARY OUTCOMES:
overall survival | 12 months
number of complete or partial responses | 6 months
  according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
worst grade toxicity per patient | evaluated every 3 weeks up to 12 months
  according to Common Toxicity Criteria for Adverse Events v. 4.03
number of patients taking oral antidiabetic therapy | at baseline
number of patients taking antithrombotic therapy | at baseline
progression free survival | 12 months
  as measured by independent central review

OTHER OUTCOMES:
predictive clinical factors for efficacy of bevacizumab | 12 months
correlation of baseline plasma biomarker expression and clinical outcome | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Nicoletta Colombo, M.D., Principal Investigator — European Institute of Oncology; Francesco Perrone, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Gennaro Daniele, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Roldano Fossati, M.D., Principal Investigator — Mario Negri Institute; Ciro Gallo, M.D., Principal Investigator — University of Campania Luigi Vanvitelli; Irene Floriani, Ph.D., Principal Investigator — Mario Negri Institute
Locations (82):
- France (29):
  - Centre Hospitalier d'Aix-en-Provence, Aix-en-Provence
  - Hôpital de la Côte Basque, Bayonne
  - Institut Bergoniè, Bordeaux
  - Hôpital Fleyriat, Bourg-en-Bresse
  - Centre François Baclesse, Caen
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre d'Oncologie et de Radiothérapie, Dijon
  - Centre Georges Francois Leclerc, Dijon
  - Centre Hospitalier du Mans, Le Mans
  - Centre Hospitalier Universitaire Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Clinique de la Sauvegarde, Lyon
  - Hôpital Nord, Marseille
  - Hôpital Saint-Joseph, Marseille
  - Clinique Claude Bernard, Metz
  - Centre Azuréen de Cancérologie, Mougins
  - Centre Hospitalier Général de Pau, Paris
  - Hopital Cochin, Paris
  - Hôpital des Diaconesses, Paris
  - Hôpital Tenon, Paris
  - Centre Hospitalier Général de Pau, Pau
  - Centre Hospitalier de la Région d'Annecy, Pringy
  - Institut Jean Godinot, Reims
  - Hopital Renè Huguenin, Institut Curie, Saint-Cloud
  - Hôpital Inter Armées de Begin (HIA Begin),, Saint-Mandé
  - GHPSO, Senlis
  - Centre de Radiothèrapie - Clinique Sainte-Anne, Strasbourg
  - Clinique des Dentellières,, Valenciennes
  - Institut de Cancérologie Gustave Roussy, Villejuif
- Greece (4):
  - Anticancer Hospital Agio Savvas, Athens
  - General Hospital of Athens Alexandra, Athens
  - General Oncology Hospital Agii Anargiri, Athens
  - General Hospital of Thessaloniki Papageorgiou, Thessaloniki
- Italy (36):
  - Centro di Riferimento Oncologico, Aviano
  - A.O. G. Rummo, Benevento
  - Spedali Civili Università di Brescia, Brescia
  - Ospedale Senatore Antonio Perrino, Brindisi
  - Fondazione del Piemonte per l'Oncologia IRCCS, Candiolo
  - Osp. Cannizzaro, Catania
  - Ospedale Civile di Faenza, Faenza
  - I.R.C.C.S. San Martino IST, Genova
  - Ospedale Galliera, Genova
  - ASL 5 Spezzino Ospedale Felettino, La Spezia
  - A.O. Vito Fazzi, Lecce
  - Ospedale Manzoni di Lecco, Lecco
  - Istituto Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori, Milan
  - U.L.S.S. 13, Mirano
  - A.O.U. Federico II, Napoli
  - A.O.U. Seconda Università di Napoli, Napoli
  - Istituto Nazionale dei Tumori , Oncologia Medica - Dipartimento Uro-Ginecologico, Napoli
  - Ist. Sacro Cuore Don Calabria, Negrar
  - NO AOU Maggiore della Carità, Novara
  - Istituto Oncologico Veneto, Padua
  - Casa di Cura La Maddalena, Palermo
  - Osp Silvestrini, Perugia
  - Ospedale Santa Chiara, Pisa
  - A.O. S. Maria degli Angeli, Pordenone
  - AO ASL 4, Prato
  - Ospedale S. Maria delle Croci AUSL di Ravenna, Ravenna
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale Civile Rimini, Rimini
  - Ospedale S. Giovanni Calibita Fatebenefratelli, Roma
  - Policlinico Universitario Gemelli Università Cattolica del Sacro Cuore, Roma
  - Policlinico Università Campus Biomedico, Roma
  - Ospedale di Sondrio, Sondrio
  - A.O. Ordine Mauriziano, Torino
  - A.O. di Udine S. Maria della Misericordia, Udine
- Centre Hospitalier Princesse Grace, Monaco, Monaco
- Switzerland (12):
  - Zentrum fùr Onkologie/ Hamat. und Transf, Aarau
  - Universitatsspital,Frauenklinik, Basel
  - IOSI, Bellinzona
  - Klinik Engeried, Bern
  - Kantonsspital, Chur
  - Kantonsspital, Frauenfeld
  - HUG Breast Center, Geneva
  - Kantonsspital, Lucerne
  - Kantonsspital, Münsterlingen
  - Kantonsspital, Olten
  - Klinische Forschung Onkologie, Sankt Gallen
  - Kantonsspital, Winterthur

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Pignata S, Lorusso D, Joly F, Gallo C, Colombo N, Sessa C, Bamias A, Salutari V, Selle F, Frezzini S, De Giorgi U, Pautier P, Bologna A, Orditura M, Dubot C, Gadducci A, Mammoliti S, Ray-Coquard I, Zafarana E, Breda E, Favier L, Ardizzoia A, Cinieri S, Largillier R, Sambataro D, Guardiola E, Lauria R, Pisano C, Raspagliesi F, Scambia G, Daniele G, Perrone F; MITO16b/MANGO-OV2/ENGOT-ov17 Investigators. Carboplatin-based doublet plus bevacizumab beyond progression versus carboplatin-based doublet alone in patients with platinum-sensitive ovarian cancer: a randomised, phase 3 trial. Lancet Oncol. 2021 Feb;22(2):267-276. doi: 10.1016/S1470-2045(20)30637-9. PMID 33539744
- [Derived] Arend R, Westin SN, Coleman RL. Decision analysis for secondline maintenance treatment of platinum sensitive recurrent ovarian cancer: a review. Int J Gynecol Cancer. 2020 May;30(5):684-694. doi: 10.1136/ijgc-2019-001041. Epub 2020 Feb 19. PMID 32079709